CLINICAL TRIAL: NCT07220265
Title: The Impact of Phenylalanine Elevations on Metabolic, Cognitive, and Neural Functioning in Adults Heterozygous for Phenylketonuria (PKU)
Brief Title: Impact of Phenylalanine Elevations on Brain and Cognition in Adult PKU Carriers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Shawn Christ, Professor, Psychological Sciences, University of Missouri-Columbia
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 2092228; R21HD115129-01A1 (NIH)
Record Dates: First submitted 2025-10-20; First posted 2025-10-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Carrier of Phenylketonuria; Healthy
MeSH Terms: interventions — Phenylalanine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PKU Carriers (Other): Heterozygous carriers of a pathogenic variant of the PAH gene associated with phenylketonuria (PKU)
  Interventions: Dietary Supplement: Phenylalanine (Phe); Dietary Supplement: Placebo
- Non-Carriers (Other): Individuals who do not carry a pathogenic variant of the PAH gene
  Interventions: Dietary Supplement: Phenylalanine (Phe); Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Phenylalanine (Phe) — Oral ingestion of phenylalanine (Phe)
Dietary Supplement: Placebo — Oral ingestion of Placebo (Vitamin C)

SUMMARY:
The goal of this clinical trial is to advance our understanding of the cognitive and neurophysiologic sequelae associated with suboptimal phenylalanine (Phe) metabolism in heterozygous carriers of phenylketonuria (PKU). The main questions it aims to answer are:

* Do PKU carriers experience prolonged elevations in brain Phe levels following oral ingestion of dietary Phe?
* Do PKU carriers experience disruptions in cognitive functioning following oral ingestion of dietary Phe?
* Do PKU carriers experience atypical brain activity following oral ingestion of dietary Phe? Researchers will compare PKU carriers and non-carriers following oral ingestion of dietary Phe and a placebo.

Participants will:

* Consume Phe or a placebo at two separate visits to our facility
* At each visit, they will complete a series of MRIs and cognitive tests throughout the day

DETAILED DESCRIPTION:
Limitations inherent in past studies of phenylketonuria (PKU) carriers (e.g., poor genetic characterization of sample resulting in inclusion of homozygous non-PKU relatives, reliance on rudimentary or overly broad behavioral assessment tools) make it difficult to conclude the extent to which neurophysiologic and cognitive processes are affected in these individuals. To address this gap in the literature, we propose to conduct a double-blind crossover study in a sample of genetically-confirmed sample of 18 heterozygous PKU carriers and 18 non-carriers. A principled investigation of the effects of elevated phenylalanine (Phe) on neurocognition will involve participants performing an fMRI n-back WM task, resting state scan, and a battery of select cognitive tests at 3 timepoints: baseline (pre-load), 2 hours and 4 hours after starting oral administration of Phe or placebo. Blood and brain levels of Phe and Tyr will also be assessed at each timepoint.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-60 years
* For the PKU carrier group: Individuals who are the parent of an individual with PKU or who are otherwise have confirmed PKU carrier status (e.g., a sibling of someone with PKU who has had genetic testing done)
* For the non-carrier group: Individuals who do not have PKU or a family history of PKU

Exclusion Criteria:

* Obesity as defined by a body mass index (BMI) over 30*
* Taking oral contraceptives on the day of testing session*
* Positive cotinine urine test showing nicotine use
* History of major neurologic condition (e.g., multiple sclerosis, severe closed head injury, Parkinson's disease)) unrelated to PKU and known to adversely impact brain health and function
* Contraindications for safe MRI participation such as (a) pregnancy or plans to become pregnant during period of study enrollment; or (b) metallic objects inside the body (e.g., surgical staples left in the body following surgery, middle ear prosthesis, metal foreign objects lodged inside the eye, heart pacemakers).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Blood Phenylalanine Levels | 3 timepoints: baseline (pre-load), 2 hours and 4 hours after starting oral administration of Phe or placebo
Brain Phenylalanine Levels | 3 timepoints: baseline (pre-load), 2 hours and 4 hours after starting oral administration of Phe or placebo
  Brain Phenylalanine Levels estimated using magnetic resonance spectroscopy (MRS)
Brain Phenylalanine-to-Tyrosine Ratio | 3 timepoints: baseline (pre-load), 2 hours and 4 hours after starting oral administration of Phe or placebo
  Ratio of Phenylalanine-to-Tyrosine concentrations in the brain as estimated using magnetic resonance spectroscopy (MRS)
Neural Activity during Go/No-Go Task | 3 timepoints: baseline (pre-load), 2 hours and 4 hours after starting oral administration of Phe or placebo
  Pattern of brain activation as captured using functional MRI while performing a go/no-go inhibitory task
Operational Span Task | 3 timepoints: baseline (pre-load), 2 hours and 4 hours after starting oral administration of Phe or placebo
  Performance-based measure of working memory ability. In this task, participants first solve a math problem and then see a letter, and then solve another math problem, and see another letter. This math-letter sequence is repeated from three to seven times for each trial with an unpredictable length each time. After each math-letter sequence, participants are asked to recall, in order, the preceding letters. Scores are calculated by summing the number of letters correctly recalled in the correct order.
Multi-Source Interference Task | 3 timepoints: baseline (pre-load), 2 hours and 4 hours after starting oral administration of Phe or placebo
  Performance-based measure of focused attention. ). In this task, participants are shown a display containing three horizontally-aligned numbers (i.e., 1, 2, or 3) and asked to respond as quickly as possible to the location (position #1, 2, or 3) of the number stimulus that is different from the others. The location may be congruent (e.g., "323") or incongruent (e.g., "112") with identity of the target number. Mean response time and error rate will served as the outcome variables.
Grooved Pegboard Test | 3 timepoints: baseline (pre-load), 2 hours and 4 hours after starting oral administration of Phe or placebo
  Performance-based measure of processing speed & fine motor control
Resting-State Functional Connectivity | 3 timepoints: baseline (pre-load), 2 hours and 4 hours after starting oral administration of Phe or placebo
  Synchronization of neural activity within brain networks as measured by functional MRI while participants are at rest

SECONDARY OUTCOMES:
Brain concentrations of glutamate, glutathione, creatine, and other metabolites | 3 timepoints: baseline (pre-load), 2 hours and 4 hours after starting oral administration of Phe or placebo
  Concentrations of various brain metabolites as estimated using magnetic resonance spectroscopy (MRS)
PROMIS Anxiety - Short Form 8a | Baseline only
  A patient-reported outcome (PRO) measure assessing symptoms of anxiety. Scores range from 8 to 40, with higher scores indicating more/worse symptoms.
PROMIS Depression - Short Form 8a | Baseline only
  A patient-reported outcome (PRO) measure assessing symptoms of depression. Scores range from 8 to 40, with higher scores indicating more/worse symptoms.
PROMIS Sleep - Short Form 8a | Baseline only
  A patient-reported outcome (PRO) measure assessing symptoms of sleep disturbance. Scores range from 8 to 40, with higher scores indicating more/worse symptoms.
PROMIS Fatigue - Short Form 8a | Baseline only
  A patient-reported outcome (PRO) measure assessing symptoms of fatigue. Scores range from 8 to 40, with higher scores indicating more/worse symptoms.
PROMIS Cognitive Function - Short Form 8a | Baseline only
  A patient-reported outcome (PRO) measure assessing symptoms of cognitive dysfunction. Scores range from 8 to 40, with higher scores indicating more/worse symptoms.
• Executive Function, Attention, and Speed Symptom Inventory (EASSI) | Baseline only
  Patient-reported outcome (PRO) measure of everyday symptoms of cognitive dysfunction. Scores range from 72 to 360, with higher scores indicating more/worse symptoms.
Adult ADHD Self-Report Scale (ASRS) | Baseline only
  Patient-reported outcome (PRO) measure of ADHD symptoms. Scores range from 0 to 124, with higher scores indicating more/worse symptoms.
Matrix Reasoning subtest from the WASI-2 | Baseline only
  Performance-based measure of fluid intelligence

CONTACTS AND LOCATIONS:
Locations (1):
- University of Missouri-Columbia, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
Demographic, blood amino acid levels, cognitive test performance, and MRI data (structural, spectroscopy, functional) will be acquired from 18 healthy adult carriers for PKU and 18 matched healthy controls. All data will be de-identified prior to deposit in the NIMH Data Archive (NDA).
Supporting Information: Study Protocol, Analytic Code
Time Frame: Data will be made available when the award ends (currently 04/30/2027)or when a publication is available, whichever comes first. As required by NDA, studies will also be created that contain the data used for every publication. Those studies will be shared when the pre-print is available. NDA will make decisions about how long to preserve the data, but that data archive has not deleted any deposited data up to now.
Access Criteria: All data will be deposited to the NDA. To request access of the data, researchers will use the standard processes at NDA, and the NDA Data Access Committee will decide which requests to grant. The standard NDA data access process allows access for one year and is renewable.